CLINICAL TRIAL: NCT01955876
Title: Drug Use Investigation of Fosrenol for Hyperphosphatemia With Chronic Kidney Disease Not on Dialysis
Brief Title: Fosrenol Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16626; FOSRENOL-PRED (Other: company internal)
Record Dates: First submitted 2013-09-06; First posted 2013-10-08 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hyperphosphatemia; Kidney Disease
Keywords: Fosrenol; hyperphosphatemia; chronic kidney disease not on dialysis
MeSH Terms: conditions — Hyperphosphatemia; Kidney Diseases | interventions — lanthanum carbonate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931)

INTERVENTIONS:
Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) — Patients treated with Fosrenol in daily clinical practice.

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan and it is a local prospective and observational study of patients who have received Fosrenol.

The objective of this research is to collect information on the safety of Fosrenol after its launching, which means collecting information on adverse events, especially adverse events in the digestive system including constipation and serious adverse events, and adverse drug reactions when the drug is administered to the below-mentioned target patients for six months.

The secondary objective is to collect information on the safety of the drug when administered for more than six months, which means collecting information on the safety of the drug when administered for up to 12 months to the target patients who have already been treated with the drug for six months. And also if at the time of 12 months after administration of Lanthanum carbonate the dialysis is not conducted, extending its' administration will be continued until conduction of dialysis, or until Sept. 30, 2015. The efficacy of fosrenol is evaluated by observing the serum P(phosphorus) level and serum PTH (parathyroid hormone) level change.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom investigators have decided to treat with Lanthanum carbonate for the first time at the respective medical institutions. Those medical institutions have to understand the objective of this investigation and conclude a written contract with Bayer Yakuhin.
* The decision to treat patients with Lanthanum carbonate will be made independently by the investigator prior to study inclusion.
* Patients treated with Lanthanum carbonate in the indication "Hyperphosphatemia" with chronic kidney disease not on dialysis".

Exclusion Criteria:

* Patients who are contraindicated based on the product label.
* Patients who have been already treated with Fosrenol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic renal failure patients who have not been treated with dialysis and will be treated with Fosrenol for hyperphosphatemia
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Incidence/number of episodes of adverse drug reactions and adverse events | 6 months after start of treatment with the drug

SECONDARY OUTCOMES:
Incidence/number of episodes of adverse drug reactions and adverse events | until the conduction of dialysis after starting the treatment with Lanthanum carbonate(Maximum 2 years)
Adverse drug event rate related to the digestive system | until the conduction of dialysis(Maximum 2 years)
Incidence/number of episodes of adverse events for 6, 12 months ,and from month 13 to the conduction of dialysis after starting the treatment with Lanthanum carbonate. | until the conduction of dialysis(Maximum 2 years)
Incidence/number of episodes of adverse drug reactions for 6, 12 months ,and from month 13 to the conduction of dialysis after starting the treatment with Lanthanum carbonate according to patient characteristics and treatment with Lanthanum carbonate. | until the conduction of dialysis(Maximum 2 years)
Serum P level for six months after start of treatment with the drug in comparison with baseline (at the time of start of treatment with fosrenol) | 6 months after start of treatment with the drug
Serum intact PTH level for six months after start of treatment with the drug in comparison with baseline | 6 months after start of treatment with the drug
Serum P level at 12 months after starting the treatment with Lanthanum carbonate in comparison with baseline (at the time of starting the treatment with Fosrenol). | 12 months
Serum P level at the conduction of dialysis from 13 months after starting the treatment with Lanthanum carbonate in comparison with baseline (at the time of starting the treatment with Fosrenol). | until the conduction of dialysis(Maximum 2 years)
Serum intact PTH level at 12 months after starting the treatment with Lanthanum carbonate in comparison with baseline (at the time of starting the treatment with Lanthanum carbonate). | 12 months
Serum intact PTH level at the conduction of dialysis from 13 months after starting the treatment with Lanthanum carbonate in comparison with baseline (at the time of starting the treatment with Lanthanum carbonate). | until the conduction of dialysis(Maximum 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan